CLINICAL TRIAL: NCT03108781
Title: The Role of Aromatherapy With Lavender Oil in the Long-term Care on a Patients Behavioral Problems Associated With Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Yan Press, Head of gariatric department, Soroka University Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SOR5244CTIL
Record Dates: First submitted 2017-03-26; First posted 2017-04-11 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2017-10

CONDITIONS: Dementia; BPSD
Keywords: Dementia; Behavioral Psychiatric symptoms; Treatment
MeSH Terms: conditions — Dementia | interventions — lavender oil; Sunflower Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lavender Oil (Active Comparator)
  Interventions: Drug: Lavender Oil; Drug: sunflower oil
- sunflower oil (Placebo Comparator)
  Interventions: Drug: Lavender Oil; Drug: sunflower oil

INTERVENTIONS:
Drug: Lavender Oil — Lavender Oil twice a day; one month on the face and one month on the legs
Drug: sunflower oil — placebo twice a day (sunflower oil); one month on the face and on month on the legs

SUMMARY:
Testing of Lavender Oil aromatherapy effect on behavior disorders in patients with severe dementia who are hospitalized in the ward for the mentally frail.

DETAILED DESCRIPTION:
Dementia as one of the most debilitating diseases presents with decline in memory and cognitive functions causing reduction in the intellectual abilities and every day functions. Today, there are estimated 24 million people suffering from dementia world wide and those numbers are expected to double every 20 years (Qiu, De Ronchi, & Fratiglioni, 2007).

About 80% of all patients suffering from dementia will develop at some point behavioural and psychological symptoms (BPSD)(Aalten et al., 2003). These symptoms will develop in at least 50% of patients treated in outpatient setting and in 75% of patients in nursing homes (Zaudig, 2000).

The behavioural and psychological symptoms (BPSD) syndrome may lead to high degree of distress in the patient and close-once, causing burnout of the primary care giver and transfer of the patient to a nursing home.

These days, the primary treatment is based on antipsychotic pharmacotherapy that is often associated with side affects and far from assured efficiency and safety (Fung, Tsang, & Chung, 2012). Research showed that the usage of antipsychotic drugs increases the chance of stroke and premature death and thus, the food and drugs administration (FDA) recommends to avoid the usage of these drugs in treatment of dementia (Ballard et al., 2009).

Non-pharmacological approach represents a good alternative in treatment of behavioural and psychological symptoms (BPSD). During the last decade the usage of alternative medicine is increasing (Fung et al., 2012), including the usage of aromatherapy in order to reduce anxiety and restlessness in dementia patients (Hersh & Falzgraf, 2007).

The treatment of behavioural and psychological symptoms (BPSD) with aromatherapy is being used for years in order to improve sleep and reduce behavioural abnormalities. However, the amount of research that studies the efficacy of aromatherapy in dementia patients is limited (Fung et al., 2012). There is lack of conclusive evidence and knowledge in the effects of dementia treatment using aromatherapy. There are two possible explanations for the conflicting and inconclusive results of studies in this area:

1. Period of treatment was too short (few minutes a day for only a week).
2. The treatment was applied far from the olfactory system (e.g., legs)

In order to confront these issues, the investigators are planning a study that will take place over the course of 4 month and will compare the treatment of aromatherapy close to the olfactory systems (i.e., face) and distant from it (i.e., legs).

ELIGIBILITY:
Inclusion Criteria:

1. Patients hospitalised in the mental frail wards of the "Mental Health Centre, Beer-Sheva".
2. Patients diagnosed with dementia (of all kinds).
3. Patients with informed consents from their guardians

Exclusion Criteria:

1. Patients without informed consent.
2. Patients with hypersensitivity to Lavender Oil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Behavioral symptoms | 4 mounths
  Behavioral symptoms will be measured by Neuropsychiatric Inventory scale

CONTACTS AND LOCATIONS:
Locations (1):
- Ben Gurion University, Beersheba, Israel

REFERENCES:
- [Derived] Ball EL, Owen-Booth B, Gray A, Shenkin SD, Hewitt J, McCleery J. Aromatherapy for dementia. Cochrane Database Syst Rev. 2020 Aug 19;8(8):CD003150. doi: 10.1002/14651858.CD003150.pub3. PMID 32813272